CLINICAL TRIAL: NCT06892080
Title: Urine Incontinence Occurrence and Sexual Hormones in Women With Chronic Spinal Cord Injury/Disease - a Pilot Study
Acronym: SexHormInkont
Status: Recruiting | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2023-15
Record Dates: First submitted 2025-03-05; First posted 2025-03-24 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injury; Urinary Incontinence; Menstrual Cycle
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premenopausal women with spinal cord injury and urinary incontinence
- Premenopausal women with spinal cord injury without urinary incontinence

SUMMARY:
There is a knowledge gap about the influence of the menstrual cycle on bladder function in women with spinal cord injury. So far, studies regarding urinary incontinence have primarily focused on women after menopause. It has become clear that a lack of the sex hormone estrogen, which occurs after menopause, can lead to urinary incontinence. During the course of the menstrual cycle, women also experience fluctuations in their sex hormones, particularly estrogen. The estrogen level is highest before ovulation and decreases afterwards. The investigators aim to explore whether this drop in hormone levels could lead to more frequent urinary incontinence during this phase. In order to offer the patients optimal treatment for urinary incontinence, it is important to understand the potential causes behind it. Participants will document their menstrual cycles and episodes of urinary incontinences over three menstrual cycles using a diary, and urine tests. This research project is a pilot study and is being conducted by Swiss Paraplegic Research at the Swiss Paraplegic Centre. The investigators are recruiting 12 participants who experience incontinence at least once a month and 12 participants who experience incontinence less frequently or not at all.

ELIGIBILITY:
Inclusion Criteria:

* women
* age ≥ 18 years
* chronic neurogenic bladder dysfunction due to acquired spinal cord injury
* regular menstrual cycle (26-30 days/cycle)
* written consent given
* UI group only: UI at least once per month

Exclusion Criteria:

* Detrusor overactivity in storage phase above 15cmH20
* Oligomenorrhea or amenorrhea (infrequent or absent menstrual periods)
* Hormonal intake/contraception
* Intake of androgens
* Intake of drugs which interfere with female sex hormones significantly
* Individuals who underwent sex reassignment surgery
* Pregnant or breastfeeding women
* Women who are trying to conceive
* Gynaecological carcinoma
* Endometriosis
* Ovariectomy
* Current pelvic floor physiotherapy
* Reconstructive surgery of bladder
* Local irritation of the bladder, such as bladder tumour, bladder stones, acute urinary tract infection at study start
* Inability to follow study procedures (cognitive or language barriers)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals with menstrual cycle
Study Population: Female outpatients of the Swiss Paraplegic Centre.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incontinence event(s) | through study completion, an average of 3 months
  Daily patient-reported events of urinary incontinence

SECONDARY OUTCOMES:
Ovulation | through study completion, an average of 3 months
  To confirm the occurrence of ovulation, urine samples are tested with luteinizing hormone (LH) stripes at following days of the menstrual cycle: 11, 12, 13, 14 and 15, where 1 is the first day of menstruation.
Recruitment rate | at study completion, an average of 2 years
  The number of eligible patients who are enrolled
Positive screening rate | at study completion, an average of 2 years
  Proportion of eligible patients who are screened
Retention rate | at study completion, an average of 2 years
  Rate of participants who finish study protocol
Assessment completion rate | at study completion, an average of 2 years
  Proportion of planned assessments that are completed
Type of urinary incontinence event | through study completion, an average of 3 months
  Daily patient-reported incontinence event: stress, urge or mixed urinary incontinence
Symptoms of urinary tract infection | through study completion, an average of 3 months
  Measured through a custom-made questionnaire at following days of the menstrual cycle: 3, 15 and 28, where 1 is the first day of menstruation.

OTHER OUTCOMES:
Maximal detrusor pressure during storage phase | Baseline
  Measured during urodynamic examination.
Bother by urinary incontinence | Baseline
  Evaluted using a numeric rating scale from 0 (no bother) to 10 (fully bothered)
Menstrual cycle anamnesis | Baseline
  Information about last menstruation, average length of the menstruation, the average length of the cycle
Bladder domain from the Australian Pelvic Floor Questionnaire | through study completion, an average of 3 months
  Impact of bladder on quality of life and overall well-being, APFQ range 0 to 48, where higher scores mean more severe symptoms: on following days of the menstrual cycle: 3, 15 and 28, where 1 is the first day of menstruation.
Bladder compliance | Baseline
  Measured during storage phase, ml/cmH2O
Bladder capacity | Baseline
  Measured during urodynamic examination.
Age | Baseline
  Time from birth to inclusion into study (years)
Date of spinal cord injury/disease onset | Baseline
Neurological level of injury | Baseline
  Highest intact spinal cord segment
ASIA score | Baseline
  The American Spinal Injury Association (ASIA) Impairment Scale (AIS) is a standardized system for assessing the severity of spinal cord injuries (SCI). It classifies the level and completeness of an injury based on motor and sensory function.
  ASIA Impairment Scale (AIS) Classification:
  A (Complete): No sensory or motor function preserved below the injury level, including the sacral segments (S4-S5).
  B (Sensory Incomplete): Sensory function preserved below the injury level, including S4-S5, but no motor function.
  C (Motor Incomplete): Some motor function preserved below the injury level, with more than half of key muscles below the level having a muscle grade <3 (not strong enough to move against gravity).
  D (Motor Incomplete): Motor function preserved below the injury level, with more than half of key muscles below the level having a muscle grade ≥3 (can move against gravity).

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Center, Nottwil, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Coded data will be shared with a gynechologist.